CLINICAL TRIAL: NCT02479984
Title: A Prospective Study Investigating the Role of Diagnostic Laparoscopy in the Preoperative Staging of Pancreatobiliary Cancer
Brief Title: Diagnostic Laparoscopy in the Preoperative Staging of Pancreatobiliary Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Sang-Jae Park, Center for Liver Cancer, National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-11-555
Record Dates: First submitted 2015-06-08; First posted 2015-06-24 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Pancreatic Cancer
Keywords: staging laparoscopy; pancreatic cancer; biliary cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Biliary Tract Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Staging laparoscopy (Experimental): Resectable pancreatobiliary cancer confirmed by radiologic studies (CT scan, MRI, PET-CT) and no evidence of distant metastasis.
  Staging laparoscopy will perform through 2 ports and a 30˚ laparoscope is inserted into the peritoneal cavity. Examining the whole abdominal wall, including the parietal and visceral peritonea, we will observe the liver surface from the dome area to the inferior surface and hepatoduodenal ligament in order to find metastatic nodules. Laparoscopic ultrasound (US) will be used to overcome in inspecting the posterior part of the liver. After complete laparoscopic examination, peritoneal lavage will be performed through the laparoscopic port.
  Interventions: Procedure: Staging Laparoscopy; Device: Laparoscopic ultrasound

INTERVENTIONS:
Procedure: Staging Laparoscopy — Resectable pancreatobiliary cancer confirmed by radiologic studies (CT scan, MRI, PET-CT) and no evidence of distant metastasis.
  Staging laparoscopy will perform through 2 ports and a 30˚ laparoscope is inserted into the peritoneal cavity. Examining the whole abdominal wall, including the parietal and visceral peritonea, we will observe the liver surface from the dome area to the inferior surface and hepatoduodenal ligament in order to find metastatic nodules. Laparoscopic ultrasound (US) will be used to overcome in inspecting the posterior part of the liver. After complete laparoscopic examination, peritoneal lavage will be performed through the laparoscopic port.
Device: Laparoscopic ultrasound

SUMMARY:
The purpose of this study is to evaluate the role of routine Staging Laparoscopy in patients with potentially resectable pancreatobiliary cancer.

DETAILED DESCRIPTION:
To evaluate the role of routine staging laparoscopy in patients with potentially resectable pancreatobiliary cancer. All analyses are performed using SAS version 9.1.3 for Windows (SAS institute, Cary, NC). Clinical and pathological variables will be analyzed using the χ2 test (or Fisher's exact test) and the Student's t test, depending on the normality of the distribution. P-values of < 0.05 are considering statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Resectable pancreatobiliary cancer confirmed by radiologic studies (CT scan, MRI, PET-CT)
2. No evidence of distant metastasis
3. aged 15-80 year old
4. performance status (PS) of 0 or 1 on Eastern Cooperative Oncology Group (ECOG) scale
5. adequate organ functions defined as indicated below

   1. WBC 3000 ~ 12 000/mm3
   2. > Hb 8.0 g/dl
   3. > Plt 100 000/mm3
   4. < Cr 1.2 mg/dl
   5. > Ccr 60 ml/min/body

Exclusion Criteria:

1. cystic neoplasm, neuroendocrine tumors
2. pregnant or breast-feeding women
3. previous upper abdominal surgery except laparoscopic cholecystectomy 4.Serious illness in medical condition

   1. unstable angina or myocardial infarction within 6 months of the trial
   2. unstable hypertension
   3. congestive heart failure
   4. severe respiratory disease requiring continuous oxygen therapy
   5. liver failure
   6. systemic administration of corticosteroids
   7. severe mental disorder

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 193 (Estimated)
Dates: Start 2011-08; Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Probability of diagnosis of metastasis (frequency) | baseline
  Probability of diagnosis of metastasis (frequency)

CONTACTS AND LOCATIONS:
Overall Officials: Sang Jae Park, MD, Principal Investigator — National Cancer Center, Korea
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea